CLINICAL TRIAL: NCT04010370
Title: Correlation of Several Formulas to Evaluate Insulin Sensitivity With the Predicted M Index (PREDIM) in Healthy Individuals
Brief Title: Correlation of Several Formulas to Evaluate Insulin Sensitivity With the Predicted M Index
Status: Completed | Type: Observational
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Manuel González Ortiz, Researcher Professor, University of Guadalajara
Other Study IDs: PREDIM-insulin sensitivity
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Results first posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Healthy Lifestyle
Keywords: Insulin sensitivity; PREDIM; Correlation; Healthy individuals
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy individuals: Cross-Sectional. No intervention. Patients of both sexes who are not sedentary or who participate in heavy physical activities and residents of the metropolitan area of Guadalajara

SUMMARY:
Recently, an index based on the oral insulin sensitivity index with glucose (OGIS) has been proposed in combination with anthropometric variables, called PREDIcted M (PREDIM), however, there is no evidence of the correlation of this with respect to the various indices (McAuley, Belfiore, Cederholm, Avignon, Matsuda, Gutt, Stumvoll, HOMA-IR (Homeostatic Model Assessment for Insulin Resistance), ISI (Insulin Sensitivity Index), Raynaud, QUICKI (The quantitative insulin sensitivity check index), FIRI (Fasting Insulin Resistance Index), Bennett, TyG (triglycerides and glucose index)) in healthy patients.

DETAILED DESCRIPTION:
Analytical cross-sectional study with 25 healthy patients of both genders (male and female) from 30 to 60 years old, residents of the metropolitan area of Guadalajara.

They will be operated on for a 3-hour oral glucose tolerance test. The insulin sensitivity will be calculated with the PREDIM, Matsuda, McAuley, Belfiore, Cederholm, Avignon, Gutt, Stumvoll, HOMA-IR, ISI, Raynaud, QUICKI, FIRI, Bennett and TyG indexes.

This protocol is already approved by the local ethics committee and written informed consent it's going to be obtained from all volunteers.

The statistical analysis will be presented with measures of central tendency and dispersion, mean and standard deviation. The nominal variables in numbers and percentages. The Kolmogorov-Smirnov test will be performed to determine if the variables follow a normal distribution. To correlate the formulas used to evaluate the insulin sensitivity with the PREDIcted M (PREDIM) technique, the Pearson or Spearman correlation will be used according to the distribution.

ELIGIBILITY:
Inclusion Criteria:

* Both genres
* Age 30 to 60 years
* BMI <25 kg / m2,
* Patients who are not sedentary or who participate in heavy physical activities
* Stable weight in the last 3 months

Exclusion Criteria:

* Blood pressure >120/80 mmHg
* Glucose >100 mg/dL
* Postprandial glucose >140 mg/dL
* Cholesterol >200 mg/dL
* Triglycerides >150 mg/dL
* Smoking
* Women with polycystic ovarian syndrome
* History of metabolic, cardiovascular, thyroid, renal, pancreatic and/or arterial hypertension
* Use of medications that modify insulin sensitivity (corticosteroids)
* Previous surgery or infection
* Symptoms of vomiting and/or excessive nausea

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients of both sexes who are not sedentary or who participate in heavy physical activities and residents of the metropolitan area of Guadalajara.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Gonzalez Ortiz, PhD, Principal Investigator — Intstituto de Terapeútica Experimental y Clínica. Universidad de Guadalajara.
Locations (1):
- Intstituto de Terapeútica Experimental y Clínica. Centro Universitario de Ciencias de la Salud. Universidad de Guadalajara, Guadalajara, Jalisco, Mexico

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Individuals: 3-hour oral glucose tolerance test (OGTT) with 75 grams of glucose load in a single time
Period: Overall Study
Arm/Group | Healthy Individuals
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Individuals
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.44 (2.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 25
Fasting glucose [Mean (Standard Deviation); unit: mmol/L] — Fasting glucose was analyzed with the glucose oxidase/peroxidase technique by enzymatic colorimetric methods on an automatic analyzer.
  mmol/L | 4.58 (0.41)
Waist circumference [Mean (Standard Deviation); unit: cm] — Waist circumference was measured with a flexible tape in the midpoint between the lowest rib and the iliac crest and is expressed in centimeters.
  cm | 78.88 (7.90)
Body weight [Mean (Standard Deviation); unit: kg] — Body weight was evaluated through a bioimpedance digital scale and results are reported in kg with a decimal.
  kg | 62.2 (9.1)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body mass index was calculated as weight (kg) divided by height (m^2).
  kg/m^2 | 22.42 (1.75)
Total cholesterol [Mean (Standard Deviation); unit: mmol/L] — Total cholesterol was analyzed with the cholesterol oxidase/peroxidase technique by enzymatic colorimetric methods on an automatic analyzer.
  mmol/L | 4.5 (0.5)
Triglycerides [Mean (Standard Deviation); unit: mmol/L] — Triglycerides were analyzed with the triglycerides oxidase/peroxidase technique by enzymatic colorimetric methods on an automatic analyzer.
  mmol/L | 0.82 (0.29)
Creatinine [Mean (Standard Deviation); unit: mmol/L] — Creatinine was analyzed with the alkaline picrate technique by enzymatic colorimetric methods on an automatic analyzer.
  mmol/L | 78.7 (23.9)
Uric acid [Mean (Standard Deviation); unit: mmol/L] — Uric acid was analyzed with the uric acid oxidase/peroxidase technique by enzymatic colorimetric methods on an automatic analyzer.
  mmol/L | 273.01 (69.59)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Blood pressure was evaluated with a digital sphygmomanometer with the subject sited down on a chair after a resting period of 5 minutes on three occasions. The mean of the three measures was considered as the value of systolic blood pressure (SBP) and diastolic (DBP).
  mmHg | 105.6 (9.72)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Blood pressure was evaluated with a digital sphygmomanometer with the subject sited down on a chair after a resting period of 5 minutes on three occasions. The mean of the three measures was considered as the value of systolic blood pressure (SBP) and diastolic (DBP).
  mmHg | 71.36 (6.53)

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity With PREDIM (PREDIcted M) Index
Description: With the results of the oral glucose tolerance test at baseline, insulin sensitivity was calculated with the PREDIM index.
  Insulin sensitivity was calculated with PREDIM index: A + B × log_e (OGIS) + C × log_e (IMC) + D × log_e (2hGlu) + log_e (INSf). A higher result is better.
  In the formula A=2.8846219; B=0.5208520; OGIS=1/2 x (B + sqrt (Bˆ2 + 4 x p5 x p6 (G120 - Gcl) x Cl OGTT)); C=-0.8223363; D=-0.4191242; E=-0.2427896; INSf=fasting insulin.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Healthy Individuals
Number analyzed (Participants) | 25
index | 72.48 (14.47)

2. Primary Outcome: Insulin Sensitivity With McAuley Index
Description: With the results of the oral glucose tolerance test at baseline, insulin sensitivity was calculated with the McAuley index.
  Insulin sensitivity was calculated with McAuley index: e[2.63-0.28 In(Insulin minute 0) - 0.31 In(Triglycerides minute 0)]. A lower result is better.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Healthy Individuals
Number analyzed (Participants) | 25
index | 46.69 (62.28)
Statistical Analysis 1: Comparison: Healthy Individuals; Correlation of McAuley index with PREDIM index at baseline; Test type: Superiority; p < 0.001, Spearman correlation

3. Primary Outcome: Insulin Sensitivity With Belfiore Index
Description: With the results of the oral glucose tolerance test at baseline, insulin sensitivity was calculated with the Belfiore index.
  Insulin sensitivity was calculated with Belfiore index: 2/((glucose minute 0/glucose minute 120) (Insulin minute 0/Insulin minute 120))+1. A higher result is better.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Healthy Individuals
Number analyzed (Participants) | 25
index | 1.52 (0.1940)
Statistical Analysis 1: Comparison: Healthy Individuals; Correlation of Belfiore index with PREDIM index at baseline; Test type: Superiority; p = 0.319, Spearman correlation

4. Primary Outcome: Insulin Sensitivity With Cederholm Index
Description: With the results of the oral glucose tolerance test at baseline, insulin sensitivity was calculated with the Cederholm index.
  Insulin sensitivity was calculated with Cederholm index: (75000+(Glucose minute 0- Glucose minute 120) x 19 x weight) / ((AUC Glucose/18) x log (AUC insulin/120)). A lower result is better.
  In the formula AUC=area under the curve.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Healthy Individuals
Number analyzed (Participants) | 25
index | 153.25 (38.93)
Statistical Analysis 1: Comparison: Healthy Individuals; Correlation of Cederholm index with PREDIM index at baseline; Test type: Superiority; p = 0.27, Spearman correlation

5. Primary Outcome: Insulin Sensitivity With Avignon Index
Description: With the results of the oral glucose tolerance test at baseline, insulin sensitivity was calculated with the Avignon index.
  Insulin sensitivity was calculated with Avignon index: ((0.137 x Sib) + Si2h)/2. A higher result is better.
  In the formula Sib=10ˆ8 / ((insulin minute 0) x (glucose minute 0) x (VD=150 ml/kg of Body weight)); Si2h=10ˆ8 / ((insulin minute 120) x (glucose minute 120) x (VD=150 ml/kg of Body weight)).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Healthy Individuals
Number analyzed (Participants) | 25
index | 271.11 (115.37)
Statistical Analysis 1: Comparison: Healthy Individuals; Correlation of Avignon index with PREDIM index at baseline; Test type: Superiority; p = 0.246, Spearman correlation

6. Primary Outcome: Insulin Sensitivity With Matsuda Index
Description: With the results of the oral glucose tolerance test at baseline, insulin sensitivity was calculated with the Matsuda index.
  Insulin sensitivity was calculated with Matsuda index: [10,000 / √glucose minute 0 x insulin minute 0) (mean glucose (OGTT) x mean insulin OGTT)]. A higher result is better.
  In the formula OGTT: oral glucose tolerance test.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Healthy Individuals
Number analyzed (Participants) | 25
index | 8.15 (3.20)
Statistical Analysis 1: Comparison: Healthy Individuals; Correlation of Matsuda index with PREDIM index at baseline; Test type: Superiority; p = 0.259, Spearman correlation

7. Primary Outcome: Insulin Sensitivity With Gutt Index
Description: With the results of the oral glucose tolerance test at baseline, insulin sensitivity was calculated with the Gutt index.
  Insulin sensitivity was calculated with Gutt index: ((75000 + (Glucose minute 0 - Glucose minute 120) x 0.10 x m) / (120 x Glucose mean x log Insulin mean). A higher result is better. A lower result is better.
  In the formula m=body weight
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Healthy Individuals
Number analyzed (Participants) | 25
index | 79.99 (16.50)
Statistical Analysis 1: Comparison: Healthy Individuals; Correlation of Gutt index with PREDIM index at baseline; Test type: Superiority; p = 0.69, Spearman correlation

8. Primary Outcome: Insulin Sensitivity With Stumvoll Index
Description: With the results of the oral glucose tolerance test at baseline, insulin sensitivity was calculated with the Stumvoll index.
  Insulin sensitivity was calculated with Stumvoll index: 0.156 - 0.0000459 × Insulin minute 120 - 0.000321 × Insulin minute 0 - 0.00541 × Glucose minute 120. A lower result is better.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Healthy Individuals
Number analyzed (Participants) | 25
index | 0.1339 (0.0242)
Statistical Analysis 1: Comparison: Healthy Individuals; Correlation of Stumvoll index with PREDIM index at baseline; Test type: Superiority; p = 0.022, Spearman correlation

9. Primary Outcome: Insulin Sensitivity With HOMA-IR (Homeostatic Model Assessment for Insulin Resistance) Index
Description: With the results of the oral glucose tolerance test at baseline, insulin sensitivity was calculated with the HOMA-IR index.
  Insulin sensitivity was calculated with HOMA-IR index: (Glucose minute 0) (Insulin minute 0) / 22.5. A lower result is better.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Healthy Individuals
Number analyzed (Participants) | 25
index | 1.61 (0.76)
Statistical Analysis 1: Comparison: Healthy Individuals; Correlation of HOMA-IR index with PREDIM index at baseline; Test type: Superiority; p = 0.69, Spearman correlation

10. Primary Outcome: Insulin Sensitivity With ISI (Insulin Sensitivity Index) Index
Description: With the results of the oral glucose tolerance test at baseline, insulin sensitivity was calculated with the ISI index.
  Insulin sensitivity was calculated with ISI index: 10000 / (Insulin minute 0) (Glucose minute 0). A lower result is better.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Healthy Individuals
Number analyzed (Participants) | 25
index | 18.61 (8.3)
Statistical Analysis 1: Comparison: Healthy Individuals; Correlation of ISI index with PREDIM index at baseline; Test type: Superiority; p = 0.69, Spearman correlation

11. Primary Outcome: Insulin Sensitivity With Raynaud Index
Description: With the results of the oral glucose tolerance test at baseline, insulin sensitivity was calculated with the Raynaud index.
  Insulin sensitivity was calculated with Raynaud index: 40 / (Fasting insulin). a lower result is better.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Healthy Individuals
Number analyzed (Participants) | 25
index | 6.05 (2.59)
Statistical Analysis 1: Comparison: Healthy Individuals; Correlation of Raynaud index with PREDIM index at baseline; Test type: Superiority; p = 0.541, Spearman correlation

12. Primary Outcome: Insulin Sensitivity With QUICKI (The Quantitative Insulin Sensitivity Check Index) Index
Description: With the results of the oral glucose tolerance test at baseline, insulin sensitivity was calculated with the QUICKI index.
  Insulin sensitivity was calculated with QUICKI index: 1 / (log fasting insulin) + (log fasting glucose). A lower result is better.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Healthy Individuals
Number analyzed (Participants) | 25
index | 0.36 (0.03)
Statistical Analysis 1: Comparison: Healthy Individuals; Correlation of QUICKI index with PREDIM index at baseline; Test type: Superiority; p = 0.69, Spearman correlation

13. Primary Outcome: Insulin Sensitivity With FIRI (Fasting Insulin Resistance Index) Index
Description: With the results of the oral glucose tolerance test at baseline, insulin sensitivity was calculated with the FIRI index.
  Insulin sensitivity was calculated with FIRI index: (Fasting Insulin) x (Fasting Glucose) / 25. A lower result is better.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Healthy Individuals
Number analyzed (Participants) | 25
index | 26.13 (12.25)
Statistical Analysis 1: Comparison: Healthy Individuals; Correlation of FIRI index with PREDIM index at baseline; Test type: Superiority; p = 0.531, Spearman correlation

14. Primary Outcome: Insulin Sensitivity With Bennett Index
Description: With the results of the oral glucose tolerance test at baseline, insulin sensitivity was calculated with the Bennett index.
  Insulin sensitivity was calculated with Bennett index: 1 / (log Fasting insulin) x (log Fasting glucose). A lower result is better.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Healthy Individuals
Number analyzed (Participants) | 25
index | 0.64 (0.15)
Statistical Analysis 1: Comparison: Healthy Individuals; Correlation of Bennett index with PREDIM index at baseline; Test type: Superiority; p = 0.726, Spearman correlation

15. Primary Outcome: Insulin Sensitivity With TyG (Triglycerides and Glucose Index) Index
Description: With the results of the oral glucose tolerance test at baseline, insulin sensitivity was calculated with the TyG index.
  Insulin sensitivity was calculated with TyG index: [ln (Triglycerides) x (Fasting Glucose) / 2]. A lower result is better.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Healthy Individuals
Number analyzed (Participants) | 25
index | 1.88 (0.08)
Statistical Analysis 1: Comparison: Healthy Individuals; Correlation of TyG index with PREDIM index at baseline; Test type: Superiority; p = 0.787, Spearman correlation

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 3 hours
Groups:
- Healthy Individuals: Subjects of both sexes (men and women), aged 30-60 years under 3-hour oral glucose tolerance test (OGTT) with 75 grams of glucose load in a single time
Arm/Group | Healthy Individuals
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT04010370/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT04010370/ICF_001.pdf